CLINICAL TRIAL: NCT03992443
Title: A Phase 3, Open Label, Single Arm Study on the Use of CUSA-081 for Dysfunctional Central Venous Access Devices (CVADs)
Brief Title: Efficacy and Safety of CUSA-081 in the Restoration of Dysfunctional Central Venous Access Device (CVAD) Functionality
Acronym: READY 2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Chiesi business decision
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUSA-081-HEM-02; 2021-004026-30 (EudraCT Number)
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Restoration of Function to CVADs
Keywords: CVAD; CUSA-081; reteplase
MeSH Terms: interventions — reteplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CUSA-081 (Experimental): Participants received 1 or 2 doses of CUSA-081, 0.70 milligrams (mg) per 2 milliliter (mL) directly into the catheter lumen. Participants received the first dose at minute (min) 0, and the second dose, if needed, at min 90. Assessments were performed at min 30, 60, 90, 120, 150, and 180.
  Interventions: Drug: CUSA-081

INTERVENTIONS:
Drug: CUSA-081 — Participants received 1 or 2 doses of CUSA-081, 0.70 mg/2 mL, directly into the catheter lumen
  Other Names: reteplase

SUMMARY:
Study to evaluate the efficacy and safety of CUSA-081 in the restoration of central venous access device (CVAD) functionality in participants 12 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. Inability to have 3 mL of blood withdrawn from the selected study catheter;
2. A single or multi-lumen CVAD, implanted ports or peripherally inserted central catheters (PICCs) in place for > 24 hours and documented as previously being patent and functional;
3. Ability to designate one dysfunctional lumen of a multi-lumen catheter to be used throughout the study for both study drug instillation and assessment of CVAD function;
4. Male and non-pregnant female subjects at least 18 years or older (see note below);
5. Able to have fluids infused at the volume necessary to instill study drug into the CVAD (i.e., up to 2 mL);
6. Informed consent form (ICF) signed and dated indicating that the subject has been informed of and agreed with all pertinent aspects of the study and is willing to comply with all study requirements and procedures.

NOTE: A urine pregnancy test is required for all females of childbearing potential. Women in natural post-menopause or permanently sterile do not need to be tested for pregnancy. Natural menopause is defined as the permanent cessation of menstrual periods, determined retrospectively after a woman has experienced 12 consecutive months of lack of menstruation (amenorrhea) without any other obvious pathological or physiological cause. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

Exclusion Criteria:

1. CVAD (any type) used for Hemodialysis;
2. CVAD known to be dysfunctional for more than 48 hours;
3. Reasonable evidence of mechanical or non-thrombotic occlusion in the selected study catheter (e.g., catheter malposition or migration, sutures, kinks, or precipitates causing obstruction), radiographic assessment is not required;
4. Known or suspected catheter-related bloodstream infection (CRBSI);
5. Use of any intravenously administered fibrinolytic agent or anticoagulant (e.g., alteplase, tenecteplase, reteplase, urokinase or heparin) within 24 hours prior to the treatment period (first instillation of study drug). Use of subcutaneous low molecular weight heparin (LMWH), unfractionated heparin (UFH) or heparinoids for prophylaxis of thromboembolic events is allowed. Furthermore, the use of oral anticoagulants is allowed.
6. Known to be at high risk for bleeding events or embolic complications in the opinion of the Investigator, or has a known condition for which bleeding constitutes a significant hazard (e.g. recent stroke, recent intracranial or intraspinal surgery or serious head trauma, intracranial neoplasm, arteriovenous malformation or aneurysm, known bleeding diathesis);
7. Uncontrolled hypertension (systolic BP ≥160 or diastolic BP ≥110 mmHg) at screening;
8. Clinically unstable in the opinion of the site investigator;
9. Known to be pregnant or breastfeeding at screening;
10. Previously treated in this study (READY 2) or in study READY 1;
11. History of allergic reaction to reteplase or vial ingredients (excipients or diluents);
12. Use of any investigational drug or experimental medical device within 28 days prior to treatment; non interventional observational study participation is allowed;
13. Not mentally, socially or otherwise able to complete the trial assessments or not likely to survive beyond 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Number Of Participants Who Experienced Severe Treatment-emergent Adverse Events (TEAEs) | Day 1 (postdose) through Day 30
  TEAEs were defined as any adverse event (AE) with a start date on or after administration of the study drug (on Day 1). A severe AE was defined as an AE that was incapacitating and required medical intervention. The number of participants who experienced 1 or more severe TEAEs after dosing on Day 1 through the Follow-up Visit (Day 30) is presented. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.

SECONDARY OUTCOMES:
Percentage Of Participants Who Had Treatment Success Following A Single Instillation Of Study Drug With A Dwell Time Up To 90 Minutes | Day 1 (up to 90 mins postdose)
  Treatment success is defined as the restoration of CVAD functionality, measured as the ability to withdraw 3 mL of blood and infuse 5 mL of saline. For this assessment, dwell time was up to 90 minutes. The percentage was calculated as the number of participants who had treatment success divided by the total number of participants in the group, multiplied by 100%.
Rate Of Recurrent Catheter Dysfunction Within 30 Days Following Treatment With Study Drug | Day 1 (postdose) up to Day 30
  The rate of recurrent catheter dysfunction is defined as re-occlusion.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (7):
  - Chiesi investigational site, San Luis Obispo, California
  - Chiesi Investigational site, Torrance, California
  - Chiesi Investigational site, Tampa, Florida
  - Chiesi investigation site, Greenville, North Carolina
  - Chiesi Investigational site, Huntersville, North Carolina
  - Chiesi Investigational site, Dayton, Ohio
  - Chiesi investigational site, Ohio City, Ohio
- Bulgaria (5):
  - Chiesi investigational site, Pleven
  - Chiesi Investigational site, Plovdiv
  - Chiesi Investigational Site, Razgrad
  - Chiesi Investigational site, Sofia
  - Chiesi Investigational site, Stara Zagora
- Hungary (3):
  - Chiesi investigational site, Budapest
  - Chiesi investigational site, Kecskemét
  - Chiesi investigational site, Székesfehérvár

IPD SHARING:
Plan to Share IPD: No